CLINICAL TRIAL: NCT01924078
Title: Capecitabine Metronomic Chemotherapy Combined With Aromatase Inhibitors in Postmenopausal Hormone-receptor-positive Breast Cancer
Brief Title: Capecitabine Metronomic Chemotherapy Plus Aromatase Inhibitor for Postmenopausal Hormone Receptor Positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guangyu Liu, Vice Director of Department of Surgical Oncology,Cancer Hospital & Institute, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Metronomic Therapy
Record Dates: First submitted 2013-08-09; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; metronomic chemotherapy; aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Aromatase Inhibitors; Letrozole; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metronomic Capecitabine and AI (Experimental): Postmenopausal Hormone receptor positive breast cancer patients who wanted to conserve breast were enrolled to receive capecitabine 500mg/tid p.o plus one of the aromatase inhibitors (AIs):Anastrozole 1mg/day p.o, and who had first line or second line Letrozole therapy failure were switched to capecitabine 500mg/tid p.o plus Exemestane 25mg/day p.o；or Exemestane therapy failure were switched to capecitabine 500mg/tid p.o plus Letrozole 2.5mg/day p.o.
  Interventions: Drug: Capecitabine; Drug: aromatase Inhibitors (AIs)

INTERVENTIONS:
Drug: Capecitabine — metronomic use: capecitabine 500mg/tid
  Other Names: Xeloda
Drug: aromatase Inhibitors (AIs) — Anastrozole 1mg/day p.o,Exemestane 25mg/day,Letrozole 2.5mg/day p.o.
  Other Names: Exmestane or Letrozol or Anastrozol

SUMMARY:
The present study is to determine the adverse effects and clinical efficacy of AI combined with Capecitabine metronomic chemotherapy in postmenopausal breast cancer patients with Estrogen receptor and/or Progestrogen receptor positive.

DETAILED DESCRIPTION:
Capecitabine (Xeloda ®) is currently the most biologically active oral fluoropyrimidine drug, and is widely used as first-line and second-line rescue therapy for advanced breast cancer ,third-generation aromatase inhibitors (AI) is the preferred adjuvant endocrine therapy for Postmenopausal hormone-sensitive breast cancer. Study showed that AI combined with metronomic chemotherapy could improve the objective response and clinical benefit in neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Hormone receptor positive;
2. previously untreated patients who do not receive hormonal therapy, or initial endocrine treatment failure or first -line endocrine treatment of relapse and metastasis failure;
3. patients who do not receive hormonal therapy must be histologically confirmed invasive ductal carcinoma, can be surgery, but must be satisfied one of the following: (1) elderly (≥70 years), or with severe heart or other systemic complications, belonging to high risk of general anesthesia, (2) have will of conserving the breast,but larger tumors (≥3cm) not suitable for breast-conserving surgery.
4. patients with metastatic breast cancer must have evaluable lesions
5. normal laboratory values:
6. informed consent (ethical approval document No. :1112105-1);
7. life expectancy of at least 3 months;
8. Postmenopausal or premenopausal with bilateral oophorectomy.

Exclusion Criteria:

1. have had radiotherapy or other local treatment for measurable lesions before the start of study received within 3 months
2. organ transplant (except for autologous or allogeneic bone marrow transplantation);
3. have evidences of central nerve system metastases or have a history of mental illness that uncontrol;
4. unable to swallow tablets, or malabsorption patients, or patients with poor upper gastrointestinal integrity;
5. unwilling or unable to comply with study protocol or unable to meet the follow up;
6. patients who researchers considered were not suitable to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
adverse events | average 10 months
  adverse events (Hand-foot syndrome,Gynecological events, blood lipids, thrombosis, cardiovascular diseases,and etc.)

SECONDARY OUTCOMES:
PFS | average 10 months
  Progression-free survival (PFS)
TTF | average 10 months
  time to treatment failure（TTF)

CONTACTS AND LOCATIONS:
Overall Officials: Guang-yu Liu, MD, Principal Investigator — Fudan University
Locations (1):
- FUSCC, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li JW, Zuo WJ, Ivanova D, Jia XQ, Lei L, Liu GY. Metronomic capecitabine combined with aromatase inhibitors for new chemoendocrine treatment of advanced breast cancer: a phase II clinical trial. Breast Cancer Res Treat. 2019 Jan;173(2):407-415. doi: 10.1007/s10549-018-5024-3. Epub 2018 Oct 25. PMID 30361875